CLINICAL TRIAL: NCT04794478
Title: Evaluation of the Safety and Effectiveness of the Dexcom Continuous Glucose Monitoring (CGM) System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL-903880
Record Dates: First submitted 2021-03-02; First posted 2021-03-12 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: All systems worn will be blinded. Sensor wear locations will be pre-assigned. All sensor insertions will be performed at the clinic by subjects and/or caregivers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CGM Users (Active Comparator): Glucose challenge during clinic sessions to assess performance of CGM compared to comparator measurement.
  Interventions: Device: Dexcom Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Dexcom Continuous Glucose Monitoring System — Dexcom Continuous Glucose Monitoring System

SUMMARY:
Evaluation of the Safety and Effectiveness of the Dexcom Glucose Monitoring (CGM) System

DETAILED DESCRIPTION:
The objective of this study is to establish performance of the Dexcom CGM System (System) in comparison to a blood glucose comparator method.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 or older
* Diagnosis of Type 1 diabetes or Type 2 diabetes
* Willing to wear the required number of Systems for the total duration of study wear
* Willing to participate in Clinic Session(s) during study wear

Exclusion Criteria:

* Presence of extensive skin changes/diseases at sensor wear site(s) that preclude wearing the sensor(s) on skin
* Known allergy to medical-grade adhesives
* Pregnancy
* Hematocrit outside specification
* ≥ 18 years of age:

  * Male: 36.0%;
  * Female: 33.0%;
* 13-17 years of age: 35.0%;
* 7 years - 12 years of age: 32.0%;
* End stage renal disease and currently managed by dialysis or anticipating initiating dialysis during the study wear period
* Required or scheduled to have a Magnetic Resonance Imaging (MRI) scan, Computed Tomography (CT) scan, or diathermy during the study wear period

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 482 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Dexcom Continuous Glucose Monitoring System Performance | 10 days
  The Dexcom Continuous Glucose Monitoring (CGM) System performance will be assessed compared to the Yellow Springs Instrument (YSI) comparator venous plasma measurements

SECONDARY OUTCOMES:
System Related Adverse Device Effects | 10 days
  The Dexcom Continuous Glucose Monitoring (CGM) System will be characterized by Adverse Device Effects experienced by study participants

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - ProSciento, Chula Vista, California
  - AMCR Institute, Escondido, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Joslin Diabetes Center, Boston, Massachusetts
  - Clinical Trials of Texas, Inc. (CTT), San Antonio, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Advanced Research, Ogden, Utah
  - UVA Center for Diabetes Technology, Charlottesville, Virginia

REFERENCES:
- [Derived] Laffel LM, Bailey TS, Christiansen MP, Reid JL, Beck SE. Accuracy of a Seventh-Generation Continuous Glucose Monitoring System in Children and Adolescents With Type 1 Diabetes. J Diabetes Sci Technol. 2023 Jul;17(4):962-967. doi: 10.1177/19322968221091816. Epub 2022 Apr 25. PMID 35466707
- [Derived] Garg SK, Kipnes M, Castorino K, Bailey TS, Akturk HK, Welsh JB, Christiansen MP, Balo AK, Brown SA, Reid JL, Beck SE. Accuracy and Safety of Dexcom G7 Continuous Glucose Monitoring in Adults with Diabetes. Diabetes Technol Ther. 2022 Jun;24(6):373-380. doi: 10.1089/dia.2022.0011. Epub 2022 Feb 21. PMID 35157505